CLINICAL TRIAL: NCT06114914
Title: TapTalkTest: Development of a Non-invasive Screening Test to Detect Risk of Alzheimer's Disease Pathology
Brief Title: TapTalkTest Project:Development of a Non-invasive Screening Test to Detect Risk of Alzheimer's Disease Pathology
Acronym: TapTalkTest
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Tasmania (Other)
Responsible Party: Principal Investigator, Jane Alty, Associate Professor, University of Tasmania
Other Study IDs: UTasmania
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease; Dementia; Movement Abnormalities; Speech Disorders
Keywords: Alzheimer's disease; Dementia; preclinical; Artificial Intelligence; Machine learning
MeSH Terms: conditions — Alzheimer Disease; Dementia; Movement Disorders; Speech Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ApoE4 genotyping - to be used as a covariate in the analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ISLAND cohort: About 1,000 participants completed hand motor and speech tests online and 150 will attend the research centre for usablity assessments
  Interventions: Diagnostic Test: Tap Talk online program
- Clinical: The new app will be tested in about 100 patients at each of the ISLAND Cognitive Clinic or the Royal Hobart Hospital
  Interventions: Diagnostic Test: Tap Talk online program

INTERVENTIONS:
Diagnostic Test: Tap Talk online program — Online hand and speech motor testing

SUMMARY:
This project aims to produce a solution for the rising incidence of dementia. This is particularly pertinent in Tasmania, Australia, with a rapidly ageing population and the oldest demographics of all Australian states. The team will develop TapTalk, a new screening test that detects risk of Alzheimer's disease (AD) pathology. TapTalk, will record a person's hand movements and speech patterns with a smartphone. Computer algorithms will learn which patterns of data are associated with AD pathology. This innovative test is based on: (i) emerging research that fine motor control required for hand and speech movements is sensitive to early AD pathology and (ii) the investigators' new machine learning methods.

DETAILED DESCRIPTION:
This project aims to produce a solution for the rising incidence of dementia. This is particularly pertinent in Tasmania, with a rapidly ageing population. The investigators' will develop TapTalk, a new screening test that detects risk of Alzheimer's disease (AD) pathology. Accounting for 70% of all dementias, the brain pathology of AD progresses silently for more than 10 years before cognitive symptoms emerge (preclinical AD). It is possible to prevent 40% of dementia by modifying risk factors such as physical inactivity and smoking. However, the lack of a cost-effective screening tool means researchers and clinicians cannot target interventions, or recruit to drug trials, in early AD. Currently, cognitive tests lack sensitivity in preclinical AD, and specialist AD biomarker tests are invasive or costly.

The investigators will address the hypothesis: "Hand-speech movement patterns will detect the risk of Alzheimer's disease pathology in research and clinical cohorts" through three aims:

1. Develop and validate analytic algorithms for TapTalk by determining which combinations of hand-speech movement data most accurately detect preclinical AD
2. Develop smartphone capability for TapTalk and determine usability and validity
3. Prospectively validate TapTalk in people who have cognitive symptoms against gold-standard clinical diagnosis of Mild Cognitive Impairment (MCI) and AD dementia

AIM 1 Problem: Identify which combination of hand-speech tests will be most discriminatory.

Method: The investigators will develop software to video-record a 2-minute oral DDK (diadochokinesis) test, where participants make speech-like sounds repetitively e.g. pa-ta-ka. We already have software to collect hand movements (see TAS Test project). The research team will invite 500 ISLAND Project participants (>50 years old) with normal cognition to compete the hand-speech tests. All participants have provided blood samples for p-tau181 levels. This new assay quantifies AD pathology (using our ultrasensitive Simoa analyser) but the practicalities and cost of accessing the highly-specialist analytic equipment limit wide accessibility. We use ptau-181 as this is a highly predictive blood biomarkers of AD risk.

Analysis: The investigators will use deep neural networks to automatically track video key points (e.g. finger/thumb tips) and audio features (e.g. pa-ta-ka). A sliding window approach extracts measures (e.g. speed/rhythm) as input data for developing an algorithm that that classifies p-tau181 levels. Outcome: TapTalk protocol and algorithm.

AIM 2 Problem: Develop smartphone capabilities and age/cognitive status cut-offs Method We will develop a smartphone app. ISLAND Project participants (CANTAB cognitive tests every 24 months in-kind) will be invited to complete TapTalk online every 12 months.

Analysis: Multi-level regression models will measure within-subject variability, and group differences on TapTalk and CANTAB at baseline, 12 and 24 months.

Outcome: An externally validated TapTalk algorithm that produces AD risk scores across age and cognitive ranges.

AIM 3 Problem: Validate TapTalk in people with cognitive symptoms. Method: The clinician researchers working at the Royal Hobart Hospital (RHH) will recruit 100 patients with cognitive symptoms (>3 months) from RHH acute medical/subacute units. The research assistant (RHHF funding requested) will complete a standard cognitive screening tool (MoCA) and smartphone TapTalk then invite patients to attend the new ISLAND cognitive clinic after discharge. This 'one-stop' interdisciplinary clinic provides bulk-billed neuropsychological and geriatrician, neurologist and physiotherapist assessments. The team will also recruit 100 consecutive patients referred to the clinic by their GPs and all patients will complete TapTalk.

Analysis: The accuracy of TapTalk and MoCA will be compared to diagnosis using ROC analysis.

Outcome: TapTalk prospectively clinically validated.

ELIGIBILITY:
AIM 1 AND AIM 2 Eligibility criteria

Inclusion Criteria:

* Adults >50 years old who are participants in the ISLAND Project and who have provided a blood sample and have normal cognition and no persistent (>3 months) cognitive symptoms will be eligible.

Exclusion Criteria:

* Impaired cognition, defined by a validated cut-off score >1.5 SD above the mean total errors adjusted for age and gender on the Paired Associates Learning sub-test of CANTAB.

AIM 3 Eligibility criteria Inclusion Criteria: >3 months of persistent cognitive symptoms (patient- or family-reported) and >50 years old.

Exclusion criteria: Acutely unwell, significant impairment of hand function, or known diagnosis of mild cognitive impairment (MCI) or dementia.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AIM 1 & AIM 2 STUDY POPULATIONS The ISLAND Project (Bartlett et al doi: 10.2196/34688) is a 10-year prospective cohort study of Tasmanians >50 years old with nested interventions to reduce dementia risk. >13,000 people have been recruited, 8,500 research participants have provided detailed demographics and health data, 3,000 have completed online CANTAB cognitive tests and 1,500 have provided blood samples. ISLAND surveys are repeated annually, and cognitive tests and blood-based biomarkers are collected every second year.
  AIM 3 STUDY POPULATION Adults aged >50 years old who are admitted to the RHH medical wards or referred by their GP to the ISLAND Cognitive clinic (Alty et al doi: 10.1002/gps.5988)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Classification accuracy for blood biomarker of Alzheimer's disease, ptau181 in adults without cognitive symptoms | 2024
  Area under a receiver operating characteristic (ROC) curve - AUC
Odds ratio of cognitive decline in adults without cognitive symptoms | 2025
  Mixed effects logistic regression will be used to estimate the odds of a participant being confirmed as 'declining' at time T2 (24 months) conditioned on TapTalk score at time T1 (12 months), where the main measure of cogitive function is the CANTAB paired associate learning (PAL) test.
Classification accuracy for prospectively predicting risk of MCI and AD in adults with cognitive symptoms | 2025
  The investigators will calculate AUC for TapTalk and MoCA. 95% confidence intervals will be obtained using bootstrapping. Covariates may include age, gender, APOE4, years of education, and handedness. The investigators will estimate cut-off scores for TapTalk and MoCA to differentiate between cognitively unimpaired vs MCI, and between cognitively unimpaired vs AD using the Youden index to optimise the trade-off between sensitivity and specificity. Classification accuracy (sensitivity and specificity) using these cut-offs will be compared using McNemar's test.

CONTACTS AND LOCATIONS:
Overall Officials: James Vickers, PhD, Study Director — University of Tasmania
Locations (1):
- University of Tasmania, Hobart, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified hand and speech motor data with comparative cognitive test scores and diagnoses.

REFERENCES:
- [Background] Alty J, Lawler K, Salmon K, McDonald S, Stuart K, Cleary A, Ma J, Rudd K, Wang X, Chiranakorn-Costa S, Collins J, Merl H, Lin X, Vickers JC. A new one-stop interdisciplinary cognitive clinic model tackles rural health inequality and halves the time to diagnosis: Benchmarked against a national dementia registry. Int J Geriatr Psychiatry. 2023 Aug;38(8):e5988. doi: 10.1002/gps.5988. PMID 37592719
- [Background] Huang G, Li R, Bai Q, Alty J. Multimodal learning of clinically accessible tests to aid diagnosis of neurodegenerative disorders: a scoping review. Health Inf Sci Syst. 2023 Jul 22;11(1):32. doi: 10.1007/s13755-023-00231-0. eCollection 2023 Dec. PMID 37489153
- [Background] Bartlett L, Bindoff A, Doherty K, Kim S, Eccleston C, Kitsos A, Roccati E, Alty J, King AE, Vickers JC. An online, public health framework supporting behaviour change to reduce dementia risk: interim results from the ISLAND study linking ageing and neurodegenerative disease. BMC Public Health. 2023 Sep 29;23(1):1886. doi: 10.1186/s12889-023-16805-2. PMID 37773122
- [Background] Alty J, Bai Q, Li R, Lawler K, St George RJ, Hill E, Bindoff A, Garg S, Wang X, Huang G, Zhang K, Rudd KD, Bartlett L, Goldberg LR, Collins JM, Hinder MR, Naismith SL, Hogg DC, King AE, Vickers JC. The TAS Test project: a prospective longitudinal validation of new online motor-cognitive tests to detect preclinical Alzheimer's disease and estimate 5-year risks of cognitive decline and dementia. BMC Neurol. 2022 Jul 18;22(1):266. doi: 10.1186/s12883-022-02772-5. PMID 35850660
- [Background] Wang X, St George RJ, Bindoff AD, Noyce AJ, Lawler K, Roccati E, Bartlett L, Tran SN, Vickers JC, Bai Q, Alty J. Estimating presymptomatic episodic memory impairment using simple hand movement tests: A cross-sectional study of a large sample of older adults. Alzheimers Dement. 2024 Jan;20(1):173-182. doi: 10.1002/alz.13401. Epub 2023 Jul 30. PMID 37519032
- [Derived] Alty J, Goldberg LR, Roccati E, Lawler K, Bai Q, Huang G, Bindoff AD, Li R, Wang X, St George RJ, Rudd K, Bartlett L, Collins JM, Aiyede M, Fernando N, Bhagwat A, Giffard J, Salmon K, McDonald S, King AE, Vickers JC. Development of a smartphone screening test for preclinical Alzheimer's disease and validation across the dementia continuum. BMC Neurol. 2024 Apr 16;24(1):127. doi: 10.1186/s12883-024-03609-z. PMID 38627686
- See also: ISLAND Project - 10-year prospective cohort study that we will recruit participants from in Aims 1 and 2 — https://island.mooc.utas.edu.au/
- See also: ISLAND Clinic - a one-stop cognitive assessment clinic that we will recruit participants from in Aim 3 — https://islandclinic.utas.edu.au/